CLINICAL TRIAL: NCT01241227
Title: Prognosis Value of Transient Elastography and Non-invasive Markers of Fibrosis in Patients With Chronic Liver Disease. A Prospective Follow-up of 4,935 Person-years
Brief Title: Prognosis Value of Transient Elastography and Non-invasive Markers of Fibrosis in Patients With Chronic Liver Disease
Acronym: PVTE
Status: Completed | Type: Observational
Sponsor: Association HGE CHU Bordeaux Sud (Other)
Responsible Party: Principal Investigator, de Ledinghen, Professor, Association HGE CHU Bordeaux Sud
Other Study IDs: HLV-0403
Record Dates: First submitted 2010-10-22; First posted 2010-11-16 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Liver Fibrosis
Keywords: liver fibrosis; survival; transient elastography
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chronic liver disease: All patients with chronic liver disease followed using FibroScan and non-invasive markers

SUMMARY:
The aim of this prospective study was to compare the 5-year prognostic value of transient elastography (TE), FibroTest (FT), APRI , FIB-4, Lok, and Child-Pugh scores for predicting survival and complications of cirrhosis in patients with chronic liver diseases.

DETAILED DESCRIPTION:
A total of 1616 patients with chronic hepatitis C was included. At 5 years, 79 patients were dead (39 liver-related deaths) and 16 patients had liver transplantation. Overall survival was 91.7% and survival without liver-related death 94.4%. Survival was significantly decreased in patients diagnosed with severe fibrosis, whatever the non-invasive method used. All these methods were able to predict a shorter survival in this large population. Patients had their prognosis decreased as liver stiffness increased. By multivariate analysis, only FibroTest > 0.74 (OR 4.41, 95%CI 1.62-12.01, p=0.004) was associated with overall survival, and liver stiffness > 9.5 kPa (OR 4.71, 95%CI 1.06-21.01, p=0.04) associated with liver-related death.

ELIGIBILITY:
Inclusion Criteria:

* chronic hepatitis C
* chronic hepatitis B
* alcoholic liver disease
* non alcoholic steatohepatitis

Exclusion Criteria:

* ascitis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We included all consecutive patients with an age over eighteen and a chronic hepatitis C of any severity. The determination of chronic hepatitis C was made using standard diagnostic criteria: serological detection of hepatitis C antibodies and positive serum HCV-RNA by PCR for more than 6 months. Exclusion criteria were chronic hepatitis B virus infection and all other causes of chronic liver disease. Patients with HIV infection were included.
Sampling Method: Non-Probability Sample
Enrollment: 1830 (Actual)
Dates: Start 2003-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 months

SECONDARY OUTCOMES:
Survival without liver complications | 3 months
Survival without liver transplantation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Julien Vergniol, MD, Principal Investigator — Association HGE CHU Bordeaux Sud; Juliette Foucher, MD, Study Chair — Association HGE CHU Bordeaux Sud; Eric Terrebonne, MD, Study Chair — Association HGE CHU Bordeaux Sud; Wassil Merrouche, Study Chair — Association HGE CHU Bordeaux Sud; Victor De Ledinghen, MD, PhD, Study Director — Association HGE CHU Bordeaux Sud; Pierre-Henri Bernard, MD, Study Chair — Association HGE CHU Bordeaux Sud; Couzigou Patrice, MD, PhD, Study Chair — Association HGE CHU Bordeaux Sud
Locations (1):
- Centre d'Investigation de la Fibrose hépatique Service Hepato-Gastroentérologie Hopital Haut-Leveque, Pessac, France

REFERENCES:
- [Derived] Vergniol J, Boursier J, Coutzac C, Bertrais S, Foucher J, Angel C, Chermak F, Hubert IF, Merrouche W, Oberti F, de Ledinghen V, Cales P. Evolution of noninvasive tests of liver fibrosis is associated with prognosis in patients with chronic hepatitis C. Hepatology. 2014 Jul;60(1):65-76. doi: 10.1002/hep.27069. PMID 24519328
- [Derived] Vergniol J, Foucher J, Terrebonne E, Bernard PH, le Bail B, Merrouche W, Couzigou P, de Ledinghen V. Noninvasive tests for fibrosis and liver stiffness predict 5-year outcomes of patients with chronic hepatitis C. Gastroenterology. 2011 Jun;140(7):1970-9, 1979.e1-3. doi: 10.1053/j.gastro.2011.02.058. Epub 2011 Mar 2. PMID 21376047